CLINICAL TRIAL: NCT06729879
Title: Effect of Yoga Eye Exercises and Musculoskeletal Physiotherapy Interventions on Presbyopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Rumeysa BARUT, Research Assistant, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GaziosmanpasaUFizyoterapi
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Presbiyopi
Keywords: Presbyopia, Yoga eye exercises, Myofascial release, Postural exercise
MeSH Terms: conditions — Presbyopia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- yoga eye exercises group (Experimental): Yoga eye exercises include eight steps. These are; closing the eyes with the palms, blinking, sideways gaze, front and sideways gaze, rotational gaze, up and down gaze, nose tip gaze, and near and far gaze. After the initial evaluation, individuals will be taught how to perform the exercises and brochures describing the exercises will be given to the individuals. It will be applied as a home-based program every day for 8 weeks.
  Interventions: Other: Yoga eye exercises group:
- myofascial release and postural correction exercises group (Active Comparator): In our study, it is planned to apply 15 minutes of myofascial release. It is planned to apply 15 minutes 3 times a week for 8 weeks.
  In our study, exercises for the neck will be applied as posture correction exercises. It will consist of a 20-30 minute program. After the first evaluation, the exercises will be done together and taught to the individuals and an exercise brochure will be given. Postural correction exercises will be done together on the treatment days when myofascial release is applied. On other days, the participant will be asked to do the postural correction exercises at home. Exercise training will be applied face to face 3 times a week for 8 weeks and as a home program on other days.
  Interventions: Other: Myofascial release-postural correction exercises group
- yoga eye exercises and myofascial release-postural correction exercises group, (Placebo Comparator): People in this group will practice yoga eye exercises individually every day for 8 weeks and will be followed up once a week. People will be given brochures for the exercises and postural correction exercises in the yoga eye exercises group. People in this group will receive myofascial release therapy 3 days a week, postural correction exercises will be done together and they will be asked to do postural correction exercises on their own on the remaining days.
  Interventions: Other: Yoga eye exercises, myofascial release-postural correction exercises group
- Control Group (Sham Comparator): The control group will not receive any intervention and will receive their first evaluation and final evaluations after 8 weeks.
  Interventions: Other: control group

INTERVENTIONS:
Other: Yoga eye exercises group: — Yoga eye exercises
  Arms: yoga eye exercises group
Other: Myofascial release-postural correction exercises group — Myofascial release-postural correction exercises
  Arms: myofascial release and postural correction exercises group
Other: Yoga eye exercises, myofascial release-postural correction exercises group — Yoga eye exercises, myofascial release-postural correction exercises group
  Arms: yoga eye exercises and myofascial release-postural correction exercises group,
Other: control group — no intervention
  Arms: Control Group

SUMMARY:
In this study, the effects of neck exercises, neck massage and yoga eye exercises on presbyopia will be examined. 52 patients diagnosed with presbyopia will be included in the study. The study is single-center and will be conducted in the Tokat Gaziosmanpaşa University Hospital, Department of Ophthalmology outpatient clinic.The study will be grouped into 4 groups. The person who agrees to participate in the study will be assigned to a group. In these groups, the first group will be subjected to eye exercises. The second group will be subjected to neck exercises and massages. The third group will be subjected to eye exercises, neck exercises and massages. The fourth group will not be subjected to any intervention. The participants in the study will be evaluated before the intervention and 8 weeks later. The doctor will conduct evaluations with an eye-related device and the physiotherapist will evaluate the questionnaire, reading speed and neck angles using the photographing method.

DETAILED DESCRIPTION:
This study will be conducted by a permanent ophthalmologist from the Department of Ophthalmology at Tokat Gaziosmanpaşa University Hospital, before and after all evaluations. The ophthalmologist will be informed about the purpose and scope of the study, and in this direction, suitable individuals will be determined according to the criteria for inclusion or exclusion during eye examinations. These individuals will be given preliminary information and those who agree to participate in the study will be included in the study.Yoga eye exercises group: Yoga eye exercises include eight steps. These are; closing the eyes with the palms, blinking, sideways gaze, front and sideways gaze, rotational gaze, up and down gaze, gaze at the tip of the nose, and near and far gaze (1).It will be implemented as a home-based program every day for 8 weeks.Myofascial release-postural correction exercise group: In our study, a 15-minute myofascial release application is planned. For more efficient suboccipital release, a 5-minute upper trapezius muscle release will be applied beforehand and a 10-minute suboccipital release will be applied (2). A 15-minute application is planned, 3 times a week for 8 weeks.Neck exercise training will be applied face to face 3 times a week for 8 weeks and as a home program on other days.Yoga eye exercises, myofascial release-postural correction exercises group: People in this group will apply yoga eye exercises individually every day for 8 weeks and will be followed up once a week. People in this group will receive myofascial release treatment 3 days a week, postural correction exercises will be done together and they will be asked to do postural correction exercises on the remaining days.Control group: The control group will not receive any intervention and will receive initial evaluations and final evaluations after 8 weeks.Assessment tools; Demographic Information Form, which includes basic information about the participants in the study, Refraction Measurement, Visual Acuity Measurement, Accommodation Amplitude Evaluation, National Eye Health Institute Visual Function Scale (NEI-VFQ 25), Craniovertebral Angle Assessment and Reading Speed assessment will be performed.

References

1. Kim SD. Effects of yogic eye exercises on eye fatigue in undergraduate nursing students. Journal of Physical Therapy Science. 2016;28(6):1813.
2. Cho SH. The effect of suboccipital muscle inhibition and posture correction exercises on chronic tension-type headaches. Journal of Back and Musculoskeletal Rehabilitation. 2021;1:1-8.

ELIGIBILITY:
Inclusion criteria Being between the ages of 40-65, Being diagnosed with presbyopia by an ophthalmologist, Having the mental capacity to understand and perform the exercises, Not having a systemic disease that prevents exercise, Agreeing to participate in the study

Exclusion Criteria; People with a history of eye surgery, People with refractive errors such as myopia, hyperopia, astigmatism, etc., People with a history of head-neck and upper extremity surgery, Being diagnosed with strabismus, Being diagnosed with glaucoma, Having a neurological problem affecting visual functions, Being diagnosed with cataract, Having a history of eye inflammation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Refraction Measurement | 8 week
  Refractive errors will be measured by the ophthalmologist using the autorefractometry method.
Craniovertebral Angle Assessment: | 8 week
  Head posture will be assessed by measuring the craniovertebral angle. The craniovertebral angle is the angle formed by the horizontal plane of the line connecting the midpoint of the ear tragus to the spinous process of C7. A decrease in the craniovertebral angle indicates an increase in the anterior tilt position of the head. The craniovertebral angle will be assessed by photographing while the patient is standing with equal weight on both feet. A photograph will be taken from 1.5 meters away from the patient's shoulder level. A marker will be attached to the spinous process of C7 and a photograph will be taken from the left shoulder level.
Visual Acuity Measurement | 8 week
  The near reading chart prepared by Eğrilmez et al. based on logarithmic order will be used. This chart is a Turkish near vision chart with 11 digits, each with a 0.1 LogMAR interval, where visual acuity can be measured from 1/10 (20/200) to 10/10 (20/20).
Evaluation of Accommodation Amplitude: | 8 week
  To evaluate the accommodation amplitude (AA), the Tonoref III autorefractometer will be used. The device measures the change in the pupil diameter from 3 to 8 mm in 1 mm increments. It also measures AA from 0 to 10 D. Only the middle area is used for accommodation. The measurement ends when there is no change in accommodation for more than 6 seconds or when the measurement time reaches 30 seconds.
National Eye Health Institute Visual Functioning Scale (NEI-VFQ 25) | 8 week
  This scale is used to assess vision-related quality of life. It consists of 3 sections with 25 questions. These sections are; general health and vision, difficulties related to activities and results of vision problems. Validity and reliability were done by Toprak et al. Scores range from 0 to 100. Increasing scores indicate an increase in vision-related quality of life.
Reading Speed Evaluation | 8 week
  In order to evaluate reading performance, participants will be asked to read a text they have never encountered before out loud for one minute and their readings will be recorded. The text will be an easy text without complex words and will be prepared using sentences with at least 2 and at most 10 words. The entire text will be written in 18-point font with 3 lines between. The total number of words read in one minute, regardless of whether they are correct or incorrect, will be considered as the reading speed .
Demographic Information Form | 8 week
  A form containing questions about the socio-demographic characteristics of the participants (age, gender, height, weight, body mass index, education status, occupation) will be applied.

IPD SHARING:
Plan to Share IPD: No
I don't understand what this topic means exactly.

REFERENCES:
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC4932063/